CLINICAL TRIAL: NCT03551899
Title: An Observational Study of Intra-operative Ventilatory Management & Post-operative Pulmonary Complications
Brief Title: Intra-operative Ventilatory Management & Post-operative Pulmonary Complications
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Jean berezian, Instructor of Anesthesia, American University of Beirut Medical Center
Other Study IDs: ANES.JB.01
Record Dates: First submitted 2018-05-08; First posted 2018-06-11 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Intra-Operative Ventilatory Management; Post-Operative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Different ventilation parameters — mode of ventilation, tidal volume per body weight and PEEP settings

SUMMARY:
Background: The list of studies with inconsistent data regarding the effect of intra-operative ventilatory management on post-operative lung injury is large. The literature is lacking data on the least injurious way of ventilating surgical patients intra-operatively. This study is necessary to support future guidelines on the practice of intra-operative mechanical ventilation.

Specific Aim: The aims of this study is first to describe intra-operative ventilatory practices at the American University of Beirut Medical Center (AUBMC), (with particular focus on the mode of ventilation, tidal volume per body weight and PEEP settings) and second, to identify the post-operative complications that could be associated with particular settings.

Methodology: This is a prospective observational study that will be conducted in the operating room at AUBMC, on patients being admitted for surgeries under general anesthesia. During the patient's stay in the hospital, targeted process (patient characteristics, surgical procedure, mechanical ventilation management, anesthesiologist characteristics) and outcomes parameters (postoperative pulmonary complications) will be collected for analysis. Patients will be monitored and followed up with intraoperatively and postoperatively.

Analysis: Different parameters and outcomes will be collected and by subgrouping the patients per their medical history statistical significance will be tested to reach a correlative analysis to the outcomes documented. Statistical comparison will be made using the ANOVA, Student's t-test, and Chi-squared test. Level of statistical significance will be considered at p<0.05. Mean age, weight, height and BMI of participants in the different groups will be calculated. ANOVA test will be performed to test statistical significance to compare the different means between different subgroups. A two sided P value of less than 0.05 was considered to be significant Significance: The literature is lacking data on the least injurious way of ventilating surgical patients intra-operatively. This study is necessary to support future guidelines on the practice of intra-operative mechanical ventilation

ELIGIBILITY:
Inclusion criteria:

1. surgeries undergone under general anesthesia
2. patients above 18 years old
3. patient able to give consent
4. American Society of Anesthesiologists (ASA) = 1 to 4

Exclusion criteria:

1. Patients unable to give consent
2. Patients below 18 years old.
3. Surgeries done under spinal anesthesia or local block or under sedation.
4. Patients admitted to Intensive care unit post-operative due to surgical complications.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Surgical patients undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Intra-operative surgical procedures | 2 hours
  Type and duration (in minutes) of the surgical procedure
Intra-operative mechanical ventilation management | 2 hours
  Ventilation mode and settings

SECONDARY OUTCOMES:
Post-operative complications that could be associated with particular settings | 1 week
  atelectasis, pneumonia, aspiration, acute respiratory distress syndrome (ARDS)

CONTACTS AND LOCATIONS:
Locations (2):
- Lebanon (2):
  - AUBMC, Beirut
  - jean Beresian, Beirut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Khatib M, Zeeni C, Shebbo FM, Karam C, Safi B, Toukhtarian A, Nafeh NA, Mkhayel S, Shadid CA, Chalhoub S, Beresian J. Intraoperative mechanical power and postoperative pulmonary complications in low-risk surgical patients: a prospective observational cohort study. BMC Anesthesiol. 2024 Feb 27;24(1):82. doi: 10.1186/s12871-024-02449-1. PMID 38413871